CLINICAL TRIAL: NCT06254469
Title: Visualizing Brain Proteinopathies Using [F-18]Flornaptitril-PET in the Prediction of Clinical Progression of Mild Cognitive Impairment With Either Suspected Chronic Traumatic Encephalopathy or Alzheimer's Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CereMark Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: CMK-0301
Record Dates: First submitted 2023-11-16; First posted 2024-02-12 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease; Chronic Traumatic Encephalopathy
MeSH Terms: conditions — Alzheimer Disease; Chronic Traumatic Encephalopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part A - Lead in (Other): Part A plans to enroll 50 participants (approximately 20 participants with mild cognitive impairment [MCI] due to suspected CTE, 20 participants with MCI due to suspected AD, and 10 age-matched healthy volunteers, whose age is within 3 years of any participants with MCI due to suspected CTE or AD in Part A).
  Interventions: Drug: [F-18]Flornaptitril
- Part B - AD (Experimental): Part B plans to enroll 90 participants with MCI due to suspected AD for primary accuracy assessments of F-18 FNT-PET imaging.
  Interventions: Drug: [F-18]Flornaptitril
- Part B - CTE (Experimental): Part B plans to enroll 90 participants with MCI due to suspected CTE from concussive and percussive injuries in approximately 1:1 ratio for primary accuracy assessments of F-18 FNT-PET imaging.
  Interventions: Drug: [F-18]Flornaptitril

INTERVENTIONS:
Drug: [F-18]Flornaptitril — All participants will receive a single dose of F-18 FNT during an imaging visit.

SUMMARY:
CMK-0301 is a multi-site, randomized clinical trial to evaluate the safety and efficacy of [F-18]Flornaptitril-PET (F-18 FNT-PET) for the prediction of clinical progression of Mild Cognitive Impairment (MCI) with either Suspected Chronic Traumatic Encephalopathy (CTE) or Alzheimer's Disease (AD).

The primary objectives of the study are to: (1) To determine the accuracy of F-18 FNT-PET in prediction of clinical decline and (2) To assess the safety and tolerability of F-18 FNT.

The secondary objectives include: (1) To demonstrate the feasibility of F-18 FNT-PET in differentiation of participants with suspected chronic traumatic encephalopathy (CTE) from those with suspected Alzheimer's disease (AD) by trained image readers, (2) To evaluate disease progression in participants with suspected CTE or AD and (3) To evaluate the correlation between F-18 FNT-PET regional and summary visual reads scan and other assessments.

ELIGIBILITY:
Inclusion Criteria:

Participants with MCI enrolling in the trial must meet all the following criteria:

1. Diagnosis of MCI due to suspected CTE, and with age >45 years, or AD, and with age >50 years at the time of the Screening Visit (see Inclusion Criteria 9) 2. Participants must have a trial partner who has frequent interaction with them (approximately >3-4 times per week), will be present for all clinic visits, and can assist in compliance with trial procedures 3. Participants, or in the Investigator's opinion, participant's legally acceptable representative, and a trial partner provide informed consent as required by IRB 4. Female participants must be either surgically sterilized or post-menopausal, defined as at least 1 year without menses as reported by the participant or have a negative serum pregnancy test 5. Willing to comply with trial procedures 6. Willing to communicate with trial personnel 7. Willing to undergo longitudinal follow-up visits at 1 and 2 years after the Imaging Visit (only for Part B) 8. CDR global score of 0.5 9. Participants with MCI due to suspected CTE must meet the diagnostic standards of possible traumatic encephalopathy syndrome as all the following criteria:

a. All of the following features are required: i) Persistence of symptoms for longer than 2 years; no other neurologic disorder that is more likely to account for all the clinical features; history of head trauma exposure, progressive course; and at least 1 supportive feature ii) History of head trauma exposure, typically associated with history of concussion, although may be limited to subconcussive trauma iii) Head trauma exposure is repetitive in nature iv) Demonstrated progressive course v) Delayed symptom onset vi) Self-report or observer report of cognitive dysfunction, confirmed with objective cognitive decline documented by results of formal neuropsychological testing. Cognitive decline typically affects more than 1 domain (neuropsychological tests, visuospatial, memory, and language) b. Only 1 of the following supportive features is required: i) Emotional dysregulation: including depression, anxiety, agitation, aggression, paranoid ideation, deterioration of interpersonal relationships, or suicidality ii) Behavioral change: including violence, poor impulse control, socially inappropriate behavior, avolition, apathy, change in personality, or comorbid substance abuse iii) Motor disturbance: including bradykinesia, tremor, rigidity, gait instability, dysarthria, dysphagia, or ataxia 9. Participants with MCI due to suspected AD must meet all the following criteria:

1. Diagnosis of MCI due to suspected AD according to workgroups of the Diagnostic Guidelines of the National Institute on Aging and Alzheimer's Association (NIA-AA)
2. Documented evidence of memory decline with gradual onset and slow progression for at least 1 year. If medically documented evidence is not available, an informant may provide confirmatory evidence
3. An MMSE-2 score of 22 to 30, inclusive, at the Screening Visit
4. Biomarker positive based on predefined plasma p-tau cutoff
5. Modified Hachinski Ischemic Score of ˂4 at the Screening Visit
6. Cognitive deficits do not occur exclusively in the context of delirium
7. Cognitive deficits are not better explained by another mental disorder (e.g., major depressive disorder, schizophrenia), or other medical condition (e.g., hypothyroidism)
8. Treated with a stable dosage regimen of acetylcholinesterase inhibitors (AchEI) and/or memantine for at least 4 months prior to the Screening Visit. Participants should be expected to remain on a stable dosage regimen of these medications for the duration of the trial. Participants who are not being treated with AchEI and/or memantine at the time of the Screening Visit due to contraindications or previous failed treatment with these medications are also eligible for inclusion, if it is expected that participants will not be treated with these medications for the duration of the trial.

Inclusion Criteria for Healthy Volunteers (Part A):

1. Medically healthy, at the age within 3 years of any participants with MCI due to suspected CTE or AD in Part A, and with no clinically relevant findings on physical examination or laboratory results
2. Participants must have a trial partner who has frequent interaction with them (approximately >3-4 times per week), will be present for all clinic visits, and can assist in compliance with trial procedures
3. No cognitive impairment based upon cognitive assessment and as evaluated by the Investigator
4. No first-degree family history of early-onset AD or other neurodegenerative diseases (prior to age 65)
5. An MMSE-2 score ≥27.

Exclusion Criteria:

1. Pregnant or breastfeeding
2. Unable to remain still for duration of imaging procedure or have an inability to tolerate neuropsychological, clinical, or PET scan studies (e.g., head tremor that may cause head motion artifact, uncontrollable psychosis, acute suicidality)
3. History of stroke, transient ischemic attack, seizures, or other condition of the head or neck within 12 months prior to the Screening Visit that, in the Investigator's opinion, might affect circulation to the head or image interpretation
4. Preexisting major neurologic or other physical illness that could confound results (e.g., multiple sclerosis, diabetes, cancer)
5. Psychiatric disorder such as mania, schizophrenia, anxiety, or depression (Geriatric Depression Scale ≥10), which in the Investigator's opinion, might interfere with completing trial procedures
6. Condition or personal circumstance that, in the Investigator's opinion, might interfere with the collection of complete, good quality data
7. History of significant prescription drug, non-prescription drug, or alcohol abuse, including but not limited to marijuana, cocaine, heroin, or derivatives
8. Previously received F-18 FNT at any time, or any other investigational product (IP) within the past 30 days
9. History of allergic reactions to albumin, or severe anemia or cardiac failure in which case the use of albumin would be medically contraindicated
10. Unstable cardiac disease or uncontrolled hypertension (systolic blood pressure [BP] >170 mmHg or diastolic BP >100 mmHg)
11. Any use of benzodiazepines within 24 hours prior to all trial visits
12. Plan to take ibuprofen or naproxen within 5 days before the PET scan
13. Received any radioactive drugs or scans within the previous month or 10 half-lives of the drug, whichever is longer, or participated in imaging or other clinical research studies that might confound trial results
14. Implants (e.g., implanted cardiac pacemakers or defibrillators, insulin pumps, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips, or other medical implants that have not been certified for MRI), a history of claustrophobia in MRI, or any contraindication for MRI
15. History of any CT/MRI finding such as mass lesions or brain infection that are unrelated to the trial
16. Participated in another clinical trial for an investigational agent (other than monoclonal antibody) and taken at least one dose of trial drug, unless confirmed as placebo, within 90 days prior to the Screening Visit. The end of a previous investigational trial is defined as the date of the last dose of trial drug
17. Monoclonal antibody treatment within the previous 180 days prior to the Screening Visit
18. Plan to receive treatment of aducanumab, lecanemab, or other potentially approved treatment options for Early AD during the trial.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of F-18 FNT-PET in prediction of clinical decline | 2 years
  The correlation between predictive development of neurodegeneration as made from F-18 FNT-PET and score change from baseline on the Clinical Dementia Rating-Sum of Boxes (CDR-SB) at the 2-year Follow-up Visit
Assessment of the safety of F-18 FNT using adverse events and serious adverse events. | 2 years
  Adverse events and serious adverse events will be monitored in patients following F-18 FNT administration.
Assessment of the safety of F-18 FNT using vital signs. | 2 years
  A patients body temperature, respiratory rate, sitting radial pulse rate, and sitting systolic and diastolic blood pressures will be monitored in patients following F-18 FNT administration.
Assessment of the safety of F-18 FNT using clinical laboratory assessments. | 2 years
  A patients complete blood count with differential, free T4 Index, Vitamin B12 serum, chemistry panel (glucose, calcium, sodium, potassium, carbon dioxide, chlorine, albumin and total protein, ALP, ALT, AST, bilirubin, BUN, creatinine), benzodiazepines, uric acid, thyroid-stimulating hormone, and cholesterol will be monitored in patients following F-18 FNT administration.
Assessment of the safety of F-18 FNT using electrocardiograms | 2 years
  12-Lead electrocardiograms (ECGs) will be performed for all participants at Screening and in-person Follow-up Visit(s). Triplicate 12-lead ECG measurements will be obtained approximately 2 minutes apart. A repeat 12-lead ECG recording may be obtained to confirm ECG findings at the discretion of the Investigator. A full assessment of the ECG will be performed including P Wave, QRS Complex, and QT Interval.
Assessment of the safety of F-18 FNT using the Suicide Behavior Questionnaire-Revised | 2 years
  The Suicide Behavior Questionnaire-Revised will be given and assessed in patients following F-18 FNT administration.

SECONDARY OUTCOMES:
Feasibility of F-18 FNT-PET to differentiate suspected CTE from suspected AD. | 2 years
  The binding patterns of F-18 FNT-PET will be assed in each patient to differentiate those patients with suspected chronic traumatic encephalopathy (CTE) from those with suspected Alzheimer's disease (AD) by trained image readers using pattern determination (for presence versus no presence of CTE or AD type pattern).
Evaluation of disease progression in participants with suspected CTE or AD using the CDR-SB at the 2-year follow-up visit. | 2 years
  The change from baseline in scores on the Clinical Dementia Rating Scale Sum of Box Scores (CDR-SB) at the 2-year follow-up visit will be used to assess the disease progression in participants with suspected CTE or AD.
Evaluation of disease progression in participants with suspected CTE or AD using the 36-Item Short Form Survey (SF-36). | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of 36-Item Short Form Survey (SF-36).
Evaluation of disease progression in participants with suspected CTE or AD using the STOP-BANG Questionnaire for Sleep Apnea. | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the STOP-BANG Questionnaire for Sleep Apnea.
Evaluation of disease progression in participants with suspected CTE or AD using the Pittsburgh Sleep Quality Index. | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the Pittsburgh Sleep Quality Index.
Evaluation of disease progression in participants with suspected CTE or AD using the Mini Mental State Examination (the 2nd edition). | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the Mini Mental State Examination (the 2nd edition).
Evaluation of disease progression in participants with suspected CTE or AD using the Modified Balance Error Scoring System. | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the Modified Balance Error Scoring System.
Evaluation of disease progression in participants with suspected CTE or AD using the Modified Balance Error Scoring System.. | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the Modified Balance Error Scoring System.
Evaluation of disease progression in participants with suspected CTE or AD using the quality of life in neurological disorders (Neuro-QOL). | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the quality of life in neurological disorders (Neuro-QOL).
Evaluation of disease progression in participants with suspected CTE or AD using the Hamilton Rating Scale for Depression (17 items). | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the Hamilton Rating Scale for Depression (17 items).
Evaluation of disease progression in participants with suspected CTE or AD using the Hamilton Anxiety Scale. | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the Hamilton Anxiety Scale
Evaluation of disease progression in participants with suspected CTE or AD using the Pfeffer Functional Activities Questionnaire. | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the Pfeffer Functional Activities Questionnaire
Evaluation of disease progression in participants with suspected CTE or AD using the Geriatric Depression Scale. | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the Geriatric Depression Scale.
Evaluation of disease progression in participants with suspected CTE or AD using the Cognitive Function Instrument. | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the Cognitive Function Instrument.
Evaluation of disease progression in participants with suspected CTE or AD using the Modified Overt Aggression Scale. | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the Modified Overt Aggression Scale.
Evaluation of disease progression in participants with suspected CTE or AD using the Wechsler Memory Scale. | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the Wechsler Memory Scale.
Evaluation of disease progression in participants with suspected CTE or AD using the Logical Memory Immediate/Delayed Recall score. | 2 years
  Wechsler Memory To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the 4th edition (WMS-IV) Logical Memory Immediate/Delayed Recall score.
Evaluation of disease progression in participants with suspected CTE or AD using the Visual Memory Index score. | 2 years
  Wechsler Memory To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the Visual Memory Index score.
Evaluation of disease progression in participants with suspected CTE or AD using the Multilingual Naming Test- 32 item version. | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the Multilingual Naming Test- 32 item version (20 minutes).
Evaluation of disease progression in participants with suspected CTE or AD using the Wechsler Adult Intelligence Scale. | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the Wechsler Adult Intelligence Scale.
Evaluation of disease progression in participants with suspected CTE or AD using the Digit Span test. | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the 4th edition (WAIS-IV) Digit Span (7 minutes).
Evaluation of disease progression in participants with suspected CTE or AD using the Animal Naming Test. | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the Animal Naming Test (3 minutes).
Evaluation of disease progression in participants with suspected CTE or AD using Trail Making Test. | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the Trail Making Test: Trails A and Trails B (6 minutes).
Evaluation of disease progression in participants with suspected CTE or AD using the Test of Memory Malingering. | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the Test of Memory Malingering (20 minutes).
Evaluation of disease progression in participants with suspected CTE or AD using the Peabody Picture Vocabulary Test. | 2 years
  To evaluate disease progression in participants with suspected CTE or AD using change from baseline of the Peabody Picture Vocabulary Test (15 minutes).
Evaluation of the correlation between F-18 FNT-PET and baseline clinical and demographic data. | 2 years
  To evaluate the correlation between F-18 FNT-PET images and a patient's baseline clinical and demographic data. The evaluation of the correlation between F-18 FNT-PET and baseline clinical and demographic data does not explicitly include the baseline clinical and demographic data.
Evaluation of the correlation between F-18 FNT-PET and conversion to dementia | 2 years
  To evaluate the correlation between F-18 FNT-PET images and a patient's conversion to dementia. The evaluation of the correlation between F-18 FNT-PET and conversion to dementia does not explicitly include the conversion to dementia data.
Evaluation of the correlation between F-18 FNT-PET and decline in executive function. | 2 years
  To evaluate the correlation between F-18 FNT-PET images and a patient's decline in executive functioning domain score of a trial specific assessment battery (neuropsychiatric and neuropsychological examinations). The evaluation of the correlation between F-18 FNT-PET and decline in executive function does not explicitly include the decline in executive function data.

OTHER OUTCOMES:
Correlation of F-18 FNT binding patterns neuropathology at autopsy. | 2 years
  To determine the correlation between regional F-18 FNT binding and regional neuropathology (concentration of tau tangles and amyloid-beta (Aβ) plaques) at autopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Chad Yucus, MD, Principal Investigator — Endeavor Health System
Locations (1):
- Endeavor Health Systems, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No